CLINICAL TRIAL: NCT05949892
Title: Efficacy of The Expanded Health Belief Model-Based Intervention in Enhancing Heart-Health Preventive Behaviors Among High School Female Students: A Randomized Controlled Trial
Brief Title: Heart-health Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mohammed Baqer Habeeb Abd Ali, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: Heart-Health Promotion
Record Dates: First submitted 2023-07-01; First posted 2023-07-18 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Heart Diseases
Keywords: Expanded Health Belief Model, Heart-Health-Preventive Behaviors, High School Female Students
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Students in the control group will be masked from any form of the proposed intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A healthy diet (Experimental): This arm will focus on the following:
  Eating lots of vegetables and fruit Choosing whole grain foods Eating protein foods Limiting highly and ultra-processed foods Highly processed foods Making water your drink of choice Salt, sodium and potassium Refraining from added sugars
  Interventions: Behavioral: Expanded Health Belief Model-Based Intervention
- Healthy Weight Management (Experimental): This arm will focus on the following:
  Physical Activity for a Healthy Weight Preventing Weight Gain Choosing an Eating Plan to Prevent Weight Gain Balancing Food and Activity for Healthy Weight
  Interventions: Behavioral: Expanded Health Belief Model-Based Intervention
- Physical Activity (Experimental): This arm will focus on the following:
  Step 1: Make a commitment Step 2: Take stock of where you are Step 3: Set realistic goals Step 4: Identify resources for information and support Step 5: Continually "check in" with yourself to monitor your progress. Revisit the goals you set for yourself in Step 3 and evaluate your progress regularly
  Interventions: Behavioral: Expanded Health Belief Model-Based Intervention
- Stress management (Experimental): This arm will focus on the following:
  Stress relief Relaxation techniques Meditation Mindfulness exercises
  Interventions: Behavioral: Expanded Health Belief Model-Based Intervention
- Smoking Cessation and Avoidance (Experimental): This arm will focus on the following:
  Second-hand smoke Offering option to avoid secondhand smoke
  Interventions: Behavioral: Expanded Health Belief Model-Based Intervention

INTERVENTIONS:
Behavioral: Expanded Health Belief Model-Based Intervention — A healthy Diet Healthy Weight Physical Activity Stress Management Smoking Cessation and Avoidance

SUMMARY:
The researchers intend to use the Expanded Health Belief Model in enhancing heart-health preventive behaviors among high school female students

DETAILED DESCRIPTION:
The study intervention will be derived from the Expanded Health Belief Model which includes adhering to healthy diet, encouraging healthy weight, nutrition, and physical activity stress management, and smoking cessation and smoking avoidance.

ELIGIBILITY:
Inclusion Criteria:

* High school female students who do not experience any psychiatric-mental disorder

Exclusion Criteria:

* High school female students who experience any psychiatric-mental disorder

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — High school female students
Enrollment: 144 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Behavioral Intention Scale for Adherence to Heart-Health Preventive Behaviors | 6 months
  Enhancing Heart-Health Preventive Behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided